CLINICAL TRIAL: NCT05683340
Title: A Placebo-controlled, Randomized, Multicenter, Double-blind, Parallel-group Trial to Confirm the Superiority of ETC-1002 in Patients With Hyper-LDL Cholesterolemia
Brief Title: A Confirmatory Trial of ETC-1002 in Patients With Hyper-LDL Cholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 346-102-00002
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Hyper-low-density Lipoprotein (LDL) Cholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETC-1002 180mg (Experimental)
  Interventions: Drug: 180mg of ETC-1002(bempedoic acid)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 180mg of ETC-1002(bempedoic acid) — 180mg, tablet, once daily, for 12 weeks
  Arms: ETC-1002 180mg
Drug: Placebo — placebo, tablet, once daily, for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the superiority of ETC-1002 after 12 weeks of administration at 180 mg/day to placebo in patients with hyper-LDL cholesterolemia who have inadequate control of low-density lipoprotein cholesterol (LDL C).

ELIGIBILITY:
Inclusion Criteria:

* Patients with inadequate response to statins or statin intolerance as defined below [Inadequate response to statins] Patients with hyper-LDL cholesterolemia who have been taking statins[and other lipid-modifying therapies(LMTs) if needed] and cannot achieve the lipid management goals of LDL-C [Statin intolerance] Patients with hyper-LDL cholesterolemia for whom safety problems have occurred while taking at least one type of statin, and who experienced resolution of the problems after discontinuation or dose reduction, and who cannot achieve the lipid management goals of LDL-C. Patients must be on the lowest or under the dosage of the approved dose of statin and/or on stable LMT(s).
* Patients with fasting TG levels of <400 mg/dL at screening
* Other protocol specific inclusion criteria may apply

Exclusion Criteria:

* Females who are pregnant or breast-feeding or who have a positive pregnancy test (urine) result at screening or baseline visits
* Patients with homozygous familial hypercholesterolemia (HoFH)
* Patients who currently have or who have had within the past 3 months prior to screening any cardiovascular diseases, or those who have developed any cardiovascular diseases during the screening or before baseline visit
* Uncontrolled hypertension, defined as sitting systolic blood pressure after resting 5 minutes of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg at screening
* Patients with uncontrolled and serious hematologic or coagulation disorders or with hemoglobin of <10.0 g/dL at screening
* Patients with uncontrolled diabetes with HbA1c of ≥9% at screening
* Patients with uncontrolled hypothyroidism with thyroid-stimulating hormone (TSH) of >1.5 × ULN at screening
* Patients with liver disease or dysfunction, including:

  * Positive serology for hepatitis B surface antigen (HBsAg) or a positive hepatitis C virus (HCV) antibody test at screening
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) of ≥3 × ULN or total bilirubin of ≥2 × ULN at screening
* Patients with creatine kinase (CK) of >3 × ULN at screening
* Patients with a history or current renal dysfunction, nephritic syndrome, or nephritis, and with estimated glomerular filtration rate (eGFR) of ≤30 mL/min/1.73 m2 at screening
* Other protocol specific exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Rinku General Medical Center, Izumisano, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: "Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Groups:
- ETC-1002 180 mg: ETC-1002 180 mg tablet once daily for 12 weeks.
- Placebo: Placebo tablet once daily for 12 weeks.
Period: Overall Study
Arm/Group | ETC-1002 180 mg | Placebo
Started | 48 | 48
Completed | 46 | 45
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETC-1002 180 mg | Placebo | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 25 | 45
  >=65 years | 28 | 23 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (13.02) | 63.9 (12.98) | 64.2 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 20 | 25 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 48 | 48 | 96
Region of Enrollment [Number; unit: participants]
  Japan | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in LDL-C From Baseline to Week 12
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week -1 and Day 1.
Time Frame: Baseline, week12
Population: The full analysis set (FAS) will include all subjects who receive at least one dose of IMP during the treatment period and for whom LDL-C values at baseline and at least one post-dose are observed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 46 | 45
Percent Change | -25.25 (1.864) | -3.46 (1.901)
Statistical Analysis 1: Comparison: ETC-1002 180 mg vs Placebo; Test type: Superiority; p = 0.001, MMRM; Least squares mean difference = -21.78, 95% CI 2-sided [-26.71 to -16.85], Standard Error of Mean 2.482 — The least squares mean difference was calculated as the value for the ETC-1002 180 mg arm minus the value for the placebo arm

2. Secondary Outcome: Percent Change in Non-HDL Cholesterol From Baseline to Week 12
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100.
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 46 | 45
Percent Change | -20.33 (1.704) | -2.76 (1.720)

3. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 46 | 45
Percent Change | -16.36 (1.405) | -2.23 (1.409)

4. Secondary Outcome: Percent Change in Apolipoprotein B From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 46 | 45
Percent Change | -18.10 (1.762) | -0.67 (1.799)

5. Secondary Outcome: Percent Change in High Sensitivity C Reactive Protein From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 46 | 45
Percent Change | 15.40 (65.246) | 119.60 (66.542)

6. Secondary Outcome: Percent Change in Hemoglobin A1c From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 46 | 45
Percent Change | -0.87 (0.590) | 0.16 (0.594)

7. Secondary Outcome: Proportion of Subjects Whose LDL-C Value Achieved the Lipid Management Goals Based on Risk Assessment at Week 12
Description: The proportion of subjects whose LDL-C value achieves the lipid management goal at Week 12.
Time Frame: Baseline, week12
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 48 | 48
Participants | 30 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up for up to 28 (+7) days after the last dose of study medication, up to 21 weeks
Description: The safety analysis set will include subjects who receive at least one dose of IMP during the treatment period.
Arm/Group | ETC-1002 180 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 13/48 | 6/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETC-1002 180 mg (N=48) | Placebo (N=48)
Nasopharyngitis (Infections and infestations) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT05683340/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT05683340/SAP_001.pdf